CLINICAL TRIAL: NCT06755099
Title: Experience of Vaginismus in Outpatient Attendants in Assiut University Women's Health Hospital: Prevalence, Impact on Quality of Life and Management
Brief Title: Female Sexual Dysfunction Assessment and Managment of Vaginismus
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa M. Mostafa, assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treatment trials in vaginismus
Record Dates: First submitted 2024-12-12; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Female Sexual Dysfunction
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- botox injection arm (Experimental): patients in this group will be treated by Botox injection
  Interventions: Drug: Botox
- radio frequency arm (Experimental): patients in this group will be treated by radio frequency
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Drug: Botox — The patient will be placed in gynecological position. Subsequently, the patient will be anesthetized with propofol bolus, a total of 270 mg IV sterilization of valval area with antiseptic solution then digital examination to assess the spasm of intriotus and vaginal walls under lowest possible doses then increasing the doses to allow for intra vaginal injection of Botox under full sedation. Pacik technique will be adopted for Botox Injection in the vagina .
  . One vial of frozen Botox 100 U will be diluted with 2 mL saline, without foaming or shaking the vial, giving a concentration of 2.5 U/0.05 mL . Using a small sized speculum and after bending the needle to 30° to facilitate injection into sub mucosal area,1 mL (50 U) of Botox will be injected into the right bulbocavernosus then into the left side .
  Arms: botox injection arm
Device: Radiofrequency — Patients will be placed in prone position. After proper disinfection, the ischial spine (IS) and insertion point of the sacrospinous ligament will be identified using fluoroscopy medial to IS. 5 ml Lidocaine 2 % will be used to apply local anesthesia to the skin at the expected entry point for the radiofrequency cannula. Then a 20 G, 10 cm long and 1 cm active tip radiofrequency cannula will be introduced gradually utilizing 2 Hz motor stimulation until pudendal nerve is identified visually by the occurrence of contraction of the external anal sphincter muscle.
  Subsequently, pulsed radiofrequency lesioning at temperature limit of 42 C will be applied bilaterally to the pudendal nerves for 240 s (2 cycles of 120 s) after applying local anesthesia using 2 cm 2% lidocaine in its vicinity.
  Arms: radio frequency arm

SUMMARY:
The study aims at :

1. The extent female sexual dysfunction problem in community through questionnaire .
2. Compare effectiveness of two treatment options for vaginismus .

DETAILED DESCRIPTION:
Female sexual dysfunction affects 41% of reproductive-age women worldwide, making it a highly prevalent medical issue. The Diagnostic and Statistical Manual of Mental Disorders (DSM) defines female sexual dysfunction (FSD) as "any sexual complaint or problem resulting from disorders of desire, arousal, orgasm, or sexual pain that causes marked distress or interpersonal difficulty". To qualify as a dysfunction, the problem must be present more than 75% of the time, for more than 6 months, causing significant distress. According to the DSM 5 (5th edition, 2013), female sexual dysfunction entails the following disorders: sexual interest / arousal disorder, female orgasmic disorder and genito-pelvic pain / penetration disorder . Sexual dysfunction has a biopsychosocial etiology, i.e. origin of the dysfunction may stem from a biological or organic condition, a psychological condition and/or asocial condition. it is usually underreported especially in conservative communities necessitating screening in different female populations .

Vaginismus is a sexual dysfunction presented as pain and fear during sexual intercourse which is caused by intermittent and unintentional spasms of the outer one-third muscles of the vagina. Negative attitude toward sex and history of sexual abuse are the predisposing factors for vaginismus which is a culture-dependent disorder. A wide range of factors from fear of pain, bleeding and panic attack to family history and valuing the hymen are among the culture-dependent agents .

Vaginismus is classified as primary, in which the woman has never experienced painless intercourse, or secondary, in which the woman has previously experienced painless intercourse but subsequently experiences dyspareunia. Secondary vaginismus may be due to physical causes such as vaginitis or trauma during childbirth, while in some cases it may be due to psychological causes, or to a combination of causes. The treatment for secondary vaginismus is the same as for primary vaginismus .

According to various potential etiologies, a multidimensional approach should be considered for treatment of vaginismus. Caregivers should take psychological, biological, emotional, and relational factors of women and their partners into account. So far , plenty of psychological, sexual and pharmacological interventions as well as cognitive and behavioral therapy, relaxation therapy and hypnotherapy have been applied for management of vaginismus which had positive effects to some extent.

Radiofrequency has been beingapplied since decades for vaginal rejuvenation and previous researches have proven the efficacy of energy-based minimally invasive radiofrequency devices for vaginal tightening . In addition, this method might offer benefits for women with genitourinary syndrome including female sexual dysfunction (FSD) and stress urinary incontinence (SUI); however, there seems to be a need for robust data and high-quality evidence. A recent study has confirmed the positive effects of temperature controlled dual-mode radiofrequency for management of vaginal laxity and improvement of pelvic floor muscles as well as female sexual function.

More recent approaches may include local injections of botulinum toxin. Type A botulinum toxin proteolytically degrades the synaptosomal-associated protein 25 (SNAP-25), a protein required for vesicle fusion and neurotransmitter release, preventing secretory vesicles from releasing the neurotransmitters, therefore blocking neuromuscular junction .

Botox, (onabotulinumtoxin A) a drug derived from a Botulinum toxin, interferes with the chemical transmitter, acetylcholine, that is responsible for muscle contraction or spasm. Botox has proven to be as safe as aspirin. It has been used for decades to weaken over-active muscles and glands in patients with conditions such as cerebral palsy, stroke , hyper hidrosis, and migraines, as well as for cosmetic purposes .

After thorough research of literature, the studies comparing Botox injection and pulsed radiofrequency in treatment of vaginismus are lacking.

ELIGIBILITY:
Inclusion Criteria:

* • Age from 18to 40 years.

  * Women diagnosed with primary vaginismus.

Vaginismus has been classified by Lamont (12) according to its severity into four degrees or grades:

1. In first degree (also known as grade 1 vaginismus), the patient has spasm of the pelvic floor that can be relieved with reassurance.
2. In the second degree, the spasm is present throughout the pelvis even with reassurance.
3. In third degree, the patient elevates her buttocks to avoid being examined.
4. In fourth degree vaginismus, the most severe form of vaginismus, the patient elevates the buttocks, retreats, and tightly closes her thighs to avoid examination

Exclusion Criteria:

* Refusing to participate in the study

  * Women whose husbands have an erectile dysfunction.
  * women with secondary vaginismus.
  * Women with psychiatric disorders.
  * Lacking the appropriate cooperation for treatment and follow-up procedure.
  * Having any contraindications to receiving botulinum, including allergies to albumin, botulinum toxin, or its injection components.
  * Previous history of treatment with botulinum or physiotherapy.
  * Infection at the injection site.
  * Diseases involving nerves and muscles, such as myasthenia gravis and Lambert-Eaton syndrome, vulvodynia, cutaneous problems at the vulva or perineum, anal fissure, urinary duct or rectum disorders, and coagulation disorders urging them to use anticoagulation drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
- prevalence of female sexual dysfunction and vaginal penetration pain disorders - prevalence of female sexual dysfunction and vaginal penetration pain disorders. | 1 year
Reevaluate female sexual function index score after intervention | 6 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- women's health hospital of Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR

REFERENCES:
- [Background] Ferreira JR, Souza RP. Botulinum toxin for vaginismus treatment. Pharmacology. 2012;89(5-6):256-9. doi: 10.1159/000337383. PMID 22507920
- [Background] Pacik PT, Geletta S. Vaginismus Treatment: Clinical Trials Follow Up 241 Patients. Sex Med. 2017 Jun;5(2):e114-e123. doi: 10.1016/j.esxm.2017.02.002. Epub 2017 Mar 28. PMID 28363809
- [Background] Matak I, Bolcskei K, Bach-Rojecky L, Helyes Z. Mechanisms of Botulinum Toxin Type A Action on Pain. Toxins (Basel). 2019 Aug 5;11(8):459. doi: 10.3390/toxins11080459. PMID 31387301
- [Background] Stachowicz AM, Hoover ML, Karram MM. Clinical utility of radiofrequency energy for female genitourinary dysfunction: past, present, and future. Int Urogynecol J. 2021 Jun;32(6):1345-1350. doi: 10.1007/s00192-021-04735-9. Epub 2021 Mar 4. PMID 33661319
- [Background] Juhasz MLW, Korta DZ, Mesinkovska NA. Vaginal Rejuvenation: A Retrospective Review of Lasers and Radiofrequency Devices. Dermatol Surg. 2021 Apr 1;47(4):489-494. doi: 10.1097/DSS.0000000000002845. PMID 33165070
- [Background] Banaei M, Kariman N, Ozgoli G, Nasiri M. Bio-psychosocial factor of vaginismus in Iranian women. Reprod Health. 2021 Oct 18;18(1):210. doi: 10.1186/s12978-021-01260-2. PMID 34663378
- [Background] Fadul R, Garcia R, Zapata-Boluda R, Aranda-Pastor C, Brotto L, Parron-Carreno T, Alarcon-Rodriguez R. Psychosocial Correlates of Vaginismus Diagnosis: A Case-Control Study. J Sex Marital Ther. 2019;45(1):73-83. doi: 10.1080/0092623X.2018.1484401. Epub 2019 Feb 7. PMID 30044690
- [Background] McCool-Myers M, Theurich M, Zuelke A, Knuettel H, Apfelbacher C. Predictors of female sexual dysfunction: a systematic review and qualitative analysis through gender inequality paradigms. BMC Womens Health. 2018 Jun 22;18(1):108. doi: 10.1186/s12905-018-0602-4. PMID 29929499